CLINICAL TRIAL: NCT02545569
Title: Evaluation of New Custom Made Hearing Product Technology and Shell Modification
Acronym: CPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Phonak AG, Switzerland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: KEK-ZH-Nr. 2014-0459
Record Dates: First submitted 2015-08-19; First posted 2015-09-10 (Estimated); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Hearing Loss, Bilateral or Unilateral
MeSH Terms: conditions — Hearing Loss | interventions — Hearing Aids

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hearing Device Type A (Active Comparator): In the ear (ITE) hearing aid, 1-3 weeks wearing
  Interventions: Device: hearing aid (MD class IIa) - ITE, BTE, RIC
- Hearing Device Type B (Experimental): In the ear (ITE) hearing aid, 1-3 weeks wearing
  Interventions: Device: hearing aid (MD class IIa) - ITE, BTE, RIC

INTERVENTIONS:
Device: hearing aid (MD class IIa) - ITE, BTE, RIC — Hearing aid means any wearable instrument or device designed for, offered for the purpose of, or represented as aiding persons with or compensating for, impaired hearing.
  Other Names: hearing accessory (MD class I) - DM systems, FM systems, remote control

SUMMARY:
The purpose of this evaluation is to receive the greatest benefit of new custom made hearing product technology and shell modification for the end customer and to continual improve the custom made hearing products.

DETAILED DESCRIPTION:
This is a controlled, single blinded comparative study which is conducted monocentric at Phonak Headquarters in Staefa.

The purpose of the studies is to evaluate the strengths and weaknesses of new custom product development in comparison to existing/old products. The results should promote the custom product development, to provide a maximum of benefit and wearing comfort to the hearing aid user.

ELIGIBILITY:
Inclusion Criteria:

* Only adult participants between 18 and 99 years
* lnformed Consent as documented by signature (Appendix lnformed Consent Form)
* Ability to fill in a questionnaire conscientious
* Healthy outer ear (w/o previous surgical procedures)

Exclusion Criteria:

* Contraindications to the MD in this study, e.g. known hypersensitivity or allergy to the investigational product,
* Limited mobility and not in the position to attend weekly appointments
* Limited ability to describe listening impressions/experiences and the use of the hearing aid
* lnability to produce a reliable hearing test result when pure tone audiometry is attempted by the audiologist
* Massively limited dexterity
* Psychological problems
* Central hearing problems

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-01-06 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Objective measurement of speech intelligibility related to the intervention. | 5 years
  SNR (speech to noise ratio) in decibel.
Objective measurement of the transfer function related to the intervention. | 5 years
  REM (real ear measurement) in decibel.
Objective measurement from the position of the outer ear related to the test subject. | 5 years
  Measurement in degree.
Objective measurement from the size of the outer ear related to the test subject. | 5 years
  Measurement in micron.
Objective measurement of humidity in the ear canal related to the test subject and the intervention. | 5 years
  Measurement in percent.
Objective measurement of temperature in the ear canal related to the test subject and the intervention. | 5 years
  Measurement in degree centigrade.

SECONDARY OUTCOMES:
Subjective rating of the intervention via questionnaire. | 5 years
  Ordinal scale

CONTACTS AND LOCATIONS:
Overall Officials: Jana-Kosima Schwarzlos, B.Sc., Principal Investigator — Switzerland, Sonova AG, CH-8712 Staefa, Zurich
Locations (1):
- Sonova AG, Stäfa, Canton of Zurich, Switzerland